CLINICAL TRIAL: NCT05426239
Title: Treatment Patterns and Outcomes in Patients With Advanced Melanoma: A Retrospective Study Using Data From the German ADOREG Registry
Brief Title: Treatment Patterns and Outcomes in Participants With Advanced Melanoma in Germany Using a German Database
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-8XH
Record Dates: First submitted 2022-06-16; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Advanced Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Participants initiating first-line systemic therapy to treat advanced melanoma.

SUMMARY:
This study is a non-interventional retrospective observational study performed on secondary data from a German multi-site cohort registry, the German national registry of skin cancer (ADOReg).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent for inclusion in ADOReg registry must be documented at study site
* Diagnosis of advanced (nonresectable or metastatic) melanoma in stage III or stage IV
* Participants received any systemic therapy to treat the advanced melanoma
* First-line systemic treatment was initiated within the index window (19-Jun-2015 to 30-Jun-2018)

Exclusion Criteria:

* Age <18 years at index date
* Receipt of clinical trial study drug at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult participants diagnosed with advanced melanoma in the ADOReg database. Participants were included based on the following:
  * a diagnosis of advanced (unresectable or metastasized) melanoma at stage III or IV according to American Joint Committee on Cancer or AJCC staging
  * Participants receive systemic therapy to treat the advanced melanoma
  * First-line treatment was initiated within the index window (19-Jun-2015 to 30-Jun-2018)
Sampling Method: Non-Probability Sample
Enrollment: 1008 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to a maximum of 4 years of follow-up

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to a maximum of 4 years of follow-up
Objective Response Rate (ORR) | Up to a maximum of 4 years of follow-up
Duration of Response (DOR) | Up to a maximum of 4 years of follow-up
Treatment-free Interval (TFI) | Up to a maximum of 4 years of follow-up
Treatment-free Survival (TFS) | Up to a maximum of 4 years of follow-up
Incidence Rate (IR) of Adverse Drug Responses (ADRs) | Up to a maximum of 4 years of follow-up
Resolution Rate (RR) of ADRs | Up to a maximum of 4 years of follow-up
Frequency of ADRs | Up to a maximum of 4 years of follow-up
Time to Treatment Discontinuation | Up to a maximum of 4 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Site0001, Frankfurt, Germany

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm